CLINICAL TRIAL: NCT02047409
Title: Prognostic Value of Oscillatory Pattern of Sympathetic Nerve Activity Muscle in Patients With Heart Failure
Brief Title: Prognostic Value of Sympathetic Modulation in Patients With Heart Failure
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: InCor Heart Institute (Other); Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Sponsor
Other Study IDs: EDT-13001-PD; 2013/07651-7 (Other: FAPESP); 2010/50048-1 (Other: FAPESP)
Record Dates: First submitted 2014-01-24; First posted 2014-01-28 (Estimated); Last update posted 2015-09-22 (Estimated); Status verified 2015-09

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to determine whether oscillatory pattern of sympathetic nerve activity muscle is an efficient index for the prognosis of patients with heart failure.

ELIGIBILITY:
Inclusion Criteria:

* Patients with systolic heart failure and New York Heart Association (NYHA)
* Ischemic, hypertensive, or idiopathic etiology
* Left ventricular ejection fraction less than 40%

Exclusion Criteria:

* Neuromuscular, Orthopedic, Neurologic and Pulmonary Diseases
* Renal failure
* Diabetes mellitus type II

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The sample consisted of patients with heart failure in clinical follow up at the Heart Institute (InCor), University of São Paulo, School of Medicine.
Sampling Method: Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2013-10; Primary Completion 2016-10 (Estimated); Study Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
Peripheral autonomic control | 12 months
  Evaluate if the reduction in the oscillatory pattern of muscle sympathetic nerve activity is associated with morbidity and mortality in patients with heart failure in a clinical follow-up 12 months

SECONDARY OUTCOMES:
Arterial baroreflex control | 12 months
Blood inflammatory markers | 12 months
Cardiac and peripheral autonomic control | 12 months
Functional Capacity | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Heart Institute (InCor), University of Sao Paulo, School of Medicine., São Paulo, São Paulo, Brazil